CLINICAL TRIAL: NCT06914362
Title: Effects of Global Postural Reeducation in Patients With Nonspecific Chronic Low Back Pain: A Randomized Controlled Study
Brief Title: Global Postural Reeducation in Nonspecific Chronic Low Back Pain
Acronym: GPR-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, Selma Bouden, assistant doctor, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR-OMG-2024-007; ECR-OMG-2024-006 (Other: Charles Nicolle Hospital)
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: low back pain; global postural reeducation; pain; mobility; function
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): Conventional reeducation included manual therapy approaches such as spinal mobilization which aims to restore joint mobility and alleviate muscular tension.
  It included also exercise therapy focusing on strengthening core muscles, improving lumbar flexibility, and enhancing posture to stabilize the spine and reduce strain on surrounding structures.
  Modalities like heat therapy, cold therapy, and transcutaneous electrical nerve stimulation (TENS) were also used to manage pain and promote muscle relaxation. Additionally, education on ergonomic principles was part of the program to adopt healthy habits and prevent recurrence of pain.
  Interventions: Procedure: conventional rehabilitation
- GPR group (Experimental): Global postural reeducation included the following GPR postures according to the Souchard approach: lying on back with the legs extended and arms folded, lying on back with the legs flexed and arms folded, lying on back with the legs extended and arms open, lying on back with the legs flexed and arms open, sitting with legs extended and standing with the back against the wall.
  Each posture was performed by the patient under the physiotherapist supervision and was held for 15 to 20 minutes.
  Besides, each patient was asked to repeat the exercises daily at home.
  Interventions: Procedure: global postural reeducation; Procedure: conventional rehabilitation

INTERVENTIONS:
Procedure: global postural reeducation — Global postural reeducation included the following GPR postures according to the Souchard approach [7]: lying on back with the legs extended and arms folded, lying on back with the legs flexed and arms folded, lying on back with the legs extended and arms open, lying on back with the legs flexed and arms open, sitting with legs extended and standing with the back against the wall.
  Each posture was performed by the patient under the physiotherapist supervision and was held for 15 to 20 minutes.
  Besides, each patient was asked to repeat the exercises daily at home.
  Arms: GPR group
Procedure: conventional rehabilitation — Conventional reeducation included manual therapy approaches such as spinal mobilization which aims to restore joint mobility and alleviate muscular tension.
  It included also exercise therapy focusing on strengthening core muscles, improving lumbar flexibility, and enhancing posture to stabilize the spine and reduce strain on surrounding structures.
  Modalities like heat therapy, cold therapy, and transcutaneous electrical nerve stimulation (TENS) were also used to manage pain and promote muscle relaxation. Additionally, education on ergonomic principles was part of the program to adopt healthy habits and prevent recurrence of pain.

SUMMARY:
The aim of this study was to compare the effectiveness of GPR associated to conventional reeducation protocol to that of the conventional reeducation protocol alone on pain, mobility, function and psychological symptoms in patients with chronic non-specific LBP.

A monocentric randomized controlled study was carried out, including patients with chronic non specific LBP, who were allocated to two groups: GPR group performed GPR associated to conventional reeducation and control group performed conventional reeducation alone. Two evaluations were performed for both groups: at baseline (T0) and at the end of the 4 weeks' sessions (T1), including pain (by Visual Analog Scale), mobility (by the Fingertip-to-floor test (FFT) and the Schober index), muscle endurance (by the Shirado and the Sorensen tests), function (by the Oswestry Disability index (ODI)) and anxiety-depressive symptoms (by the Hospital Anxiety and Depression (HAD)).

DETAILED DESCRIPTION:
The aim of this study was to compare the effectiveness of GPR associated to conventional reeducation protocol to that of the conventional reeducation protocol alone on pain, mobility, function and psychological symptoms in patients with chronic non-specific LBP.

A monocentric randomized controlled trial was carried out between march and september 2024, in the department of physiotherapy and rheumatology of Charles Nicolle Hospital in Tunis, Tunisia.

The study population included patients aged 18 or older, diagnosed by a rheumatologist with chronic (≥ 12 months) non-specific LBP.

Exclusion criteria were acute and sub-acute LBP, neurological complications (motor impairment and cauda equina syndrome), specific causes of LBP (such as tumors, chronic rheumatic diseases infections and vertebral fracture) and pregnancy. Patients who had received other physiotherapeutic interventions or undergone surgical spinal procedures within 6 months prior to the baseline assessment were also excluded.

The included patients were allocated to two groups: GPR group performed GPR associated to conventional reeducation and control group performed conventional reeducation alone.

All patients gave their written consent before being included in the study. The study was approved by the local ethics committee of our hospital according to the number FWA00032745.

Two qualified physiotherapists, with at least 5-years' experience delivered the rehabilitation program either GPR or conventional reeducation according to group assignment.

For both groups, the programs started immediately after baseline evaluation. Both programs lasted 12 sessions over a period of 4 weeks, at a frequency of 3 times per week. Each session lasted 60 minutes. All sessions were performed in the morning and were undergone by the same physiotherapist who had experience with the GPR approach.

Conventional reeducation included manual therapy approaches such as spinal mobilization which aims to restore joint mobility and alleviate muscular tension.

It included also exercise therapy focusing on strengthening core muscles, improving lumbar flexibility, and enhancing posture to stabilize the spine and reduce strain on surrounding structures.

Modalities like heat therapy, cold therapy, and transcutaneous electrical nerve stimulation (TENS) were also used to manage pain and promote muscle relaxation. Additionally, education on ergonomic principles was part of the program to adopt healthy habits and prevent recurrence of pain.

Global postural reeducation included the following GPR postures according to the Souchard approach: lying on back with the legs extended and arms folded, lying on back with the legs flexed and arms folded, lying on back with the legs extended and arms open, lying on back with the legs flexed and arms open, sitting with legs extended and standing with the back against the wall.

Each posture was performed by the patient under the physiotherapist supervision and was held for 15 to 20 minutes.

Besides, each patient was asked to repeat the exercises daily at home. Two evaluations were performed for both groups: one at baseline (T0) and one at the end of the 4 weeks' sessions (T1).

Baseline assessment concerned sociodemographic characteristics (age, gender, body mass index (BMI), profession, physical activity) and disease characteristics (disease duration).

Outcome measurements at T0 and T1 included:

* Pain, which was evaluated using the visual analog scale (VAS) of pain
* Mobility of the lumbar spine, which was evaluated with the Fingertip-to-floor test (FFT) and the Schober index.
* Muscle endurance was evaluated using the Shirado and the Sorensen tests for abdominal and spinal musculature respectively.
* Function capacity, which was assessed by the Oswestry Disability index (ODI)
* Anxiety-depressive symptoms, which were assessed by the Hospital Anxiety and Depression (HAD) scale.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or older
* diagnosed with chronic (≥ 12 months) non-specific LBP

Exclusion Criteria:

* acute and sub-acute LBP
* neurological complications (motor impairment and cauda equina syndrome)
* specific causes of LBP (such as tumors, chronic rheumatic diseases infections and vertebral fracture)
* surgical spinal procedures within 6 months
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
pain intensity | Two evaluations were performed for both groups: one at baseline (T0) and one at the end of the 4 weeks' sessions (T1).
  Pain, which was evaluated using the visual analog scale (VAS) of pain, ranging from 0 (painless) to 10 (severe pain)

SECONDARY OUTCOMES:
mobility | Two evaluations were performed for both groups: one at baseline (T0) and one at the end of the 4 weeks' sessions (T1).
  Mobility of the lumbar spine, which was evaluated the Schober index.
muscle endurance | Two evaluations were performed for both groups: one at baseline (T0) and one at the end of the 4 weeks' sessions (T1).
  Muscle endurance was evaluated using the Shirado test for abdominal and spinal musculature respectively
function | Two evaluations were performed for both groups: one at baseline (T0) and one at the end of the 4 weeks' sessions (T1).
  Function capacity, which was assessed by the Oswestry Disability index (ODI) in its Arabic version, which is structured in 10 sections aligning with various daily activities with each section scored on a six-point scale (0-5). Scores of 0-20% indicate minimal disability, 20-40% moderate disability, 40-60% severe disability, 60-80% significant impairment, 80-100% confinement to bed or potential exaggeration of symptoms.
anxiety and depression | Two evaluations were performed for both groups: one at baseline (T0) and one at the end of the 4 weeks' sessions (T1).
  Anxiety-depressive symptoms, which were assessed by the Hospital Anxiety and Depression (HAD) scale in its Arabic version. The HAD questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Nicolle Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No